CLINICAL TRIAL: NCT02997176
Title: A PHASE I OPEN-LABEL PHARMACOKINETICS AND SAFETY STUDY OF TALAZOPARIB (MDV3800) IN PATIENTS WITH ADVANCED SOLID TUMORS AND NORMAL OR VARYING DEGREES OF HEPATIC IMPAIRMENT
Brief Title: An Open-Label Pharmacokinetics and Safety Study of Talazoparib (MDV3800)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Medivation, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MDV3800-02; C3441002 (Other: Alias Study Number)
Record Dates: First submitted 2016-12-15; First posted 2016-12-19 (Estimated); Results first posted 2021-02-25 (Actual); Last update posted 2021-02-25 (Actual); Status verified 2021-02

CONDITIONS: Advanced Solid Tumors
MeSH Terms: interventions — talazoparib

ARMS (4):
- Group A (control, normal hepatic function) (Experimental)
  Interventions: Drug: Talazoparib
- Group B (mild hepatic dysfunction) (Experimental)
  Interventions: Drug: Talazoparib
- Group C (moderate hepatic dysfunction) (Experimental)
  Interventions: Drug: Talazoparib
- Group D (severe hepatic dysfunction) (Experimental)
  Interventions: Drug: Talazoparib

INTERVENTIONS:
Drug: Talazoparib — Daily oral doses of talazoparib 0.5 mg
  Other Names: MDV3800; BMN673

SUMMARY:
This is a trial to investigate the pharmacokinetics (PK) and the safety of talazoparib in patients with advanced solid tumors and impaired hepatic function.

DETAILED DESCRIPTION:
At the end of the study, patients with no clinically significant toxicities, no contraindications to continue treatment with talazoparib, and no disease progression (underlying cancer progression) may be eligible to continue talazoparib treatment in a separate open-label extension study. The decision to allow the patient to continue dosing with talazoparib in an open-label extension (OLE) study will be based on potential overall benefit-risk and patient meeting eligibility criteria for OLE.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated Informed Consent Form (by the patient or a legally acceptable representative as per the local regulations).
2. Female or male at least 18 years of age.
3. Histologically or cytologically confirmed advanced solid tumor with no available standard treatment options in the opinion of the Investigator
4. Eastern Cooperative Oncology Group (ECOG) Performance status ≤ 2.
5. Expected life expectancy of ≥ 3 months.
6. Able to swallow the study drug (no contraindication to oral agents).
7. Hepatic function at screening and enrollment as defined by the NCI organ dysfunction working group (NCI-ODWG) criteria.
8. Adequate other organ function at screening and enrollment.
9. Female patients of childbearing potential must have a negative serum pregnancy test at screening and must agree to use a highly effective form of contraception from the time of the first dose of study drug through 7 months after the last dose of study drug.
10. Male patients must agree to use a condom when having sex with a pregnant woman or with a non-pregnant female partner of childbearing potential, from 21 days before the first dose of study drug through 4 months after last dose of study drug.
11. Female patients must not be breastfeeding at screening nor during the study participation until 7 months after the last dose of the study drug.
12. Willingness and ability to comply with scheduled visits, treatment plan, laboratory tests, and other trial procedures.

Exclusion Criteria:

1. Treatment within 14 days or five half lives prior to enrollment whichever is longer with any type of systemic anticancer-therapy or any investigational drug
2. Have not recovered (recovery is defined as CTCAE grade ≤ 1) from the acute toxicities of previous anticancer standard or investigational therapy, except treatment-related alopecia or laboratory abnormalities otherwise meeting eligibility requirements.
3. Major surgery within 28 days prior to enrollment.
4. Serious accompanying cardiac disorder
5. Active known or suspected brain metastasis or active leptomeningeal disease needing treatment
6. Symptomatic or impending spinal cord compression or cauda equine syndrome
7. Has undergone a liver transplant, kidney transplant or nephrectomy.
8. Prior allergic reaction or severe intolerance (meeting the criteria for a serious adverse event, a grade 3 or 4 AE, or permanent treatment discontinuation) to a poly ADP ribose polymerase (PARP) inhibitor.
9. Known myelodysplastic syndrome
10. Seropositive for human immunodeficiency virus (HIV).
11. Any serious or unstable medical condition that interferes with ability to tolerate treatment or assessments associated with the protocol.
12. Gastrointestinal disorder affecting absorption.
13. Known or suspected hypersensitivity to any of the talazoparib capsule components.
14. Any condition or reason that interferes with ability to participate in the study, tolerate treatment or assessments associated with the protocol, causes undue risk, or complicates the interpretation of safety data, in the opinion of the Investigator or Medical Monitor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2016-09-30 (Actual); Primary Completion 2020-02-12 (Actual); Study Completion 2020-02-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (11):
- United States (11):
  - UCLA Hematology/Oncology - Alhambra, Alhambra, California
  - CBCC Global Research, Inc. at Comprehensive Blood and Cancer Center, Bakersfield, California
  - St. Joseph Heritage Healthcare, Fullerton, California
  - St. Jude Hospital Yorba Linda DBA St. Joseph Heritage Healthcare, Fullerton, California
  - UCLA Hematology/Oncology, Los Angeles, California
  - UCLA Hematology/Oncology - Porter Ranch, Porter Ranch, California
  - UCLA Hematology/Oncology - Santa Monica, Santa Monica, California
  - UCLA Torrance Oncology, Torrance, California
  - UCLA Hematology/Oncology - Santa Clarita, Valencia, California
  - Orlando Health, Inc., Orlando, Florida
  - The University of Texas MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=MDV3800-02

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants with advanced solid tumors and impaired hepatic function were enrolled. Participants were assigned to 1 of the 4 groups based on their hepatic function as per the national cancer institute organ dysfunction working group (NCI-ODWG) classification.
Groups:
- Talazoparib: Normal Hepatic Function: Participants with total bilirubin (TB) and aspartate aminotransferase (AST) less than or equal to (<=) upper limit of normal (ULN), received talazoparib 0.5 milligram (mg) (2 capsules of 0.25 mg), orally once daily for 22 days.
- Talazoparib: Mild Hepatic Impairment: Participants with TB <=ULN and AST greater than (>) ULN or TB >1.0 to 1.5* ULN and any AST value, received talazoparib 0.5 mg (2 capsules of 0.25 mg), orally once daily for 22 days.
- Talazoparib: Moderate Hepatic Impairment: Participants with TB >1.5 to 3.0 *ULN and any AST value received talazoparib 0.5 mg (2 capsules of 0.25 mg), orally once daily for 22 days.
- Talazoparib: Severe Hepatic Impairment: Participants with TB >3*ULN and any AST value received talazoparib 0.5 mg (2 capsules of 0.25 mg), orally once daily for 22 days.
Period: Overall Study
Arm/Group | Talazoparib: Normal Hepatic Function | Talazoparib: Mild Hepatic Impairment | Talazoparib: Moderate Hepatic Impairment | Talazoparib: Severe Hepatic Impairment
Started | 7 | 10 | 5 | 16
Completed | 6 | 8 | 3 | 5
Not Completed | 1 | 2 | 2 | 11
Not completed — Adverse Event | 0 | 0 | 0 | 8
Not completed — Progressive Disease | 1 | 0 | 1 | 1
Not completed — Death | 0 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 2 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all participants who received any amount of talazoparib.
Groups:
- Talazoparib: Normal Hepatic Function: Participants with TB and AST <=ULN received 0.5 mg (2 capsules of 0.25 mg) of talazoparib daily, orally for 22 days.
- Total: Total of all reporting groups
Arm/Group | Talazoparib: Normal Hepatic Function | Talazoparib: Mild Hepatic Impairment | Talazoparib: Moderate Hepatic Impairment | Talazoparib: Severe Hepatic Impairment | Total
Number analyzed (Participants) | 7 | 10 | 5 | 16 | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.3 (7.61) | 56.6 (17.08) | 60.4 (6.31) | 52.7 (11.98) | 56.1 (12.40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 7 | 5 | 9 | 26
  Male | 2 | 3 | 0 | 7 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 2 | 1 | 6
  Not Hispanic or Latino | 4 | 7 | 3 | 14 | 28
  Unknown or Not Reported | 2 | 1 | 0 | 1 | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1 | 2 | 0 | 1 | 4
  White | 5 | 8 | 5 | 13 | 31
  Other | 1 | 0 | 0 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Free Plasma Concentration Time Curve From Zero to 24 Hours (AUC0-24) of Talazoparib on Day 22
Description: AUC0-24 of talazoparib was defined as the area under the free plasma concentration time curve from time 0 to 24 hours post-dose.
Time Frame: Pre-dose (24 hours +/- 60 minutes from the previous dose on Day 21 but within 60 minutes prior to next dose), 0.5, 1, 2, 4, 6, anytime from 8 to 12 and 24 hours post-dose on Day 22
Population: Pharmacokinetic (PK) evaluable analysis population included all enrolled participants who completed Day 22 visit, missed less than 5 consecutive doses, received at least 10 consecutive days of 0.5 mg talazoparib daily dose immediately preceding Day 22 visit without dose interruption, not vomited talazoparib dose on Day 1 and last day of dose, at least 85% of total plasma PK samples collection was reported and provided at least 1 of talazoparib PK parameters of primary interest from Day 22 visit.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter
Arm/Group | Talazoparib: Normal Hepatic Function | Talazoparib: Mild Hepatic Impairment | Talazoparib: Moderate Hepatic Impairment | Talazoparib: Severe Hepatic Impairment
Number analyzed (Participants) | 6 | 6 | 3 | 2
nanogram*hour per milliliter | 111.8 (30) | 159.0 (99) | 123.6 (30) | NA (NA) — Data is not reported, as it was planned to report statistics when there were >=3 evaluable participants.
Statistical Analysis 1: Comparison: Talazoparib: Normal Hepatic Function vs Talazoparib: Mild Hepatic Impairment; AUC0-24 was natural log-transformed and analyzed using an analysis of variance (ANOVA) model with hepatic function group as a fixed effect; Test type: Other — Bioequivalence; Percent Ratio of Geometric Means = 142.19, 90% CI 2-sided [79.92 to 252.98]
Statistical Analysis 2: Comparison: Talazoparib: Normal Hepatic Function vs Talazoparib: Moderate Hepatic Impairment; [analysis description as in outcome 1, analysis 1]; Test type: Other — Bioequivalence; Percent Ratio of Geometric Means = 110.54, 90% CI 2-sided [54.58 to 223.85]

2. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of Talazoparib on Day 22
Description: Cmax was defined as the maximum observed plasma concentration of talazoparib.
Time Frame: as for outcome 1
Population: PK evaluable analysis population included all enrolled participants who completed Day 22 visit, missed less than 5 consecutive doses, received at least 10 consecutive days of 0.5 mg talazoparib daily dose immediately preceding Day 22 visit without dose interruption, not vomited talazoparib dose on Day 1 and last day of dose, at least 85% of total plasma PK samples collection was reported and provided at least 1 of talazoparib PK parameters of primary interest from Day 22 visit.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter
Arm/Group | Talazoparib: Normal Hepatic Function | Talazoparib: Mild Hepatic Impairment | Talazoparib: Moderate Hepatic Impairment | Talazoparib: Severe Hepatic Impairment
Number analyzed (Participants) | 6 | 6 | 3 | 2
nanogram per milliliter | 10.30 (23) | 11.30 (65) | 13.56 (23) | NA (NA) — Data is not reported, as it was planned to report statistics when there were >=3 evaluable participants.
Statistical Analysis 1: Comparison: Talazoparib: Normal Hepatic Function vs Talazoparib: Mild Hepatic Impairment; Cmax was natural log-transformed and analyzed using an ANOVA model with hepatic function group as a fixed effect; Test type: Other — Bioequivalence; Percent Ratio of Geometric Means = 109.76, 90% CI 2-sided [70.93 to 169.84]
Statistical Analysis 2: Comparison: Talazoparib: Normal Hepatic Function vs Talazoparib: Moderate Hepatic Impairment; Cmax was natural log-transformed and analyzed using an ANOVA model with hepatic function group as a fixed effect; Test type: Other — Bioequivalence; Percent Ratio of Geometric Means = 131.67, 90% CI 2-sided [77.14 to 224.74]

3. Primary Outcome: Unbound Area Under the Free Plasma Concentration Time Curve From Zero to 24 Hours (AUC0-24u) of Talazoparib on Day 22
Description: AUC0-24u for unbound talazoparib was defined as the area under the free plasma concentration time curve from time 0 to 24 hours post-dose. AUC0-24u = fu*AUC0-24. fu= Fraction of Unbound (fu) Plasma.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter
Arm/Group | Talazoparib: Normal Hepatic Function | Talazoparib: Mild Hepatic Impairment | Talazoparib: Moderate Hepatic Impairment | Talazoparib: Severe Hepatic Impairment
Number analyzed (Participants) | 6 | 6 | 3 | 2
nanogram*hour per milliliter | 30.17 (11) | 45.08 (84) | 33.50 (35) | NA (NA) — Data is not reported, as it was planned to report statistics when there were >=3 evaluable participants.
Statistical Analysis 1: Comparison: Talazoparib: Normal Hepatic Function vs Talazoparib: Mild Hepatic Impairment; AUC0-24u was natural log-transformed and analyzed using an ANOVA model with hepatic function group as a fixed effect; Test type: Other — Bioequivalence; Percent Ratio of Geometric Means = 149.39, 90% CI 2-sided [91.49 to 243.93]
Statistical Analysis 2: Comparison: Talazoparib: Normal Hepatic Function vs Talazoparib: Moderate Hepatic Impairment; AUC0-24u was natural log-transformed and analyzed using an ANOVA model with hepatic function group as a fixed effect; Test type: Other — Bioequivalence; Percent Ratio of Geometric Means = 111.04, 90% CI 2-sided [60.91 to 202.43]

4. Primary Outcome: Unbound Maximum Observed Plasma Concentration (Cmaxu) of Talazoparib on Day 22
Description: Cmaxu was defined as the maximum observed plasma concentration for unbound talazoparib. Cmaxu = fu*Cmax.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter
Arm/Group | Talazoparib: Normal Hepatic Function | Talazoparib: Mild Hepatic Impairment | Talazoparib: Moderate Hepatic Impairment | Talazoparib: Severe Hepatic Impairment
Number analyzed (Participants) | 6 | 6 | 3 | 2
nanogram per milliliter | 2.778 (27) | 3.204 (56) | 3.675 (28) | NA (NA) — Data is not reported, as it was planned to report statistics when there were >=3 evaluable participants.
Statistical Analysis 1: Comparison: Talazoparib: Normal Hepatic Function vs Talazoparib: Mild Hepatic Impairment; Cmaxu was natural log-transformed and analyzed using an ANOVA model with hepatic function group as a fixed effect; Test type: Other — Bioequivalence; Percent Ratio of Geometric Means = 115.32, 90% CI 2-sided [77.95 to 170.6]
Statistical Analysis 2: Comparison: Talazoparib: Normal Hepatic Function vs Talazoparib: Moderate Hepatic Impairment; Cmaxu was natural log-transformed and analyzed using an ANOVA model with hepatic function group as a fixed effect; Test type: Other — Bioequivalence; Percent Ratio of Geometric Means = 132.26, 90% CI 2-sided [81.87 to 213.67]

5. Secondary Outcome: Area Under the Free Plasma Concentration Time Curve From Zero to 24 Hours (AUC0-24) of Talazoparib on Day 1
Description: as for outcome 1
Time Frame: Pre-dose (within 60 minutes prior to dose), 0.5, 1, 2, 4, 6, anytime between 8 to 12 and 24 hours post-dose on Day 1
Population: PK parameter analysis population included all enrolled participants who received at least 1 dose of talazoparib and had at least 1 of the talazoparib PK parameters. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter
Arm/Group | Talazoparib: Normal Hepatic Function | Talazoparib: Mild Hepatic Impairment | Talazoparib: Moderate Hepatic Impairment | Talazoparib: Severe Hepatic Impairment
Number analyzed (Participants) | 7 | 8 | 5 | 13
nanogram*hour per milliliter | 22.21 (41) | 27.63 (38) | 25.20 (7) | 21.26 (58)
Statistical Analysis 1: Comparison: Talazoparib: Normal Hepatic Function vs Talazoparib: Mild Hepatic Impairment; AUC0-24 was natural log-transformed and analyzed using an ANOVA model with hepatic function group as a fixed effect; Test type: Other — Bioequivalence; Percent Ratio of Geometric Means = 124.40, 90% CI 2-sided [85.19 to 181.66]
Statistical Analysis 2: Comparison: Talazoparib: Normal Hepatic Function vs Talazoparib: Moderate Hepatic Impairment; AUC0-24 was natural log-transformed and analyzed using an ANOVA model with hepatic function group as a fixed effect; Test type: Other — Bioequivalence; Percent Ratio of Geometric Means = 113.42, 90% CI 2-sided [73.90 to 174.07]
Statistical Analysis 3: Comparison: Talazoparib: Normal Hepatic Function vs Talazoparib: Severe Hepatic Impairment; AUC0-24 was natural log-transformed and analyzed using an ANOVA model with hepatic function group as a fixed effect; Test type: Other — Bioequivalence; Percent Ratio of Geometric Means = 95.68, 90% CI 2-sided [67.90 to 134.83]

6. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Talazoparib on Day 1
Description: Cmax was defined as the maximum observed plasma concentration of talazoparib.
Time Frame: Pre-dose (within 60 minutes prior to dose), 0.5, 1, 2, 4, 6, anytime between 8 to 12 and 24 hours post-dose on Day 1
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter
Arm/Group | Talazoparib: Normal Hepatic Function | Talazoparib: Mild Hepatic Impairment | Talazoparib: Moderate Hepatic Impairment | Talazoparib: Severe Hepatic Impairment
Number analyzed (Participants) | 7 | 8 | 5 | 15
nanogram per milliliter | 3.068 (66) | 3.047 (32) | 2.959 (44) | 1.965 (90)
Statistical Analysis 1: Comparison: Talazoparib: Normal Hepatic Function vs Talazoparib: Mild Hepatic Impairment; Cmax was natural log-transformed and analyzed using an ANOVA model with hepatic function group as a fixed effect; Test type: Other — Bioequivalence; Percent Ratio of Geometric Means = 99.31, 90% CI 2-sided [57.74 to 170.80]
Statistical Analysis 2: Comparison: Talazoparib: Normal Hepatic Function vs Talazoparib: Moderate Hepatic Impairment; Cmax was natural log-transformed and analyzed using an ANOVA model with hepatic function group as a fixed effect; Test type: Other — Bioequivalence; Percent Ratio of Geometric Means = 96.45, 90% CI 2-sided [52.22 to 178.14]
Statistical Analysis 3: Comparison: Talazoparib: Normal Hepatic Function vs Talazoparib: Severe Hepatic Impairment; Cmax was natural log-transformed and analyzed using ANOVA model with hepatic function group as a fixed effect; Test type: Other — Bioequivalence; Percent Ratio of Geometric Means = 64.05, 90% CI 2-sided [39.65 to 103.46]

7. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) of Talazoparib on Day 1
Description: Tmax was defined as the time to reach maximum observed plasma concentration of talazoparib.
Time Frame: Pre-dose (within 60 minutes prior to dose), 0.5, 1, 2, 4, 6, anytime between 8 to 12 and 24 hours post-dose on Day 1
Population: as for outcome 5
Measure: Median (Full Range); unit: hour
Arm/Group | Talazoparib: Normal Hepatic Function | Talazoparib: Mild Hepatic Impairment | Talazoparib: Moderate Hepatic Impairment | Talazoparib: Severe Hepatic Impairment
Number analyzed (Participants) | 7 | 8 | 5 | 15
hour | 1.00 [0.50 to 1.02] | 1.51 [0.50 to 2.05] | 0.55 [0.48 to 1.02] | 1.00 [0.50 to 24.62]

8. Secondary Outcome: Fraction of Unbound (fu) Plasma Talazoparib on Day 1
Description: Fraction of unbound drug (fu) was defined as the ratio of unbound drug concentration to the total drug concentration and reported as percentage (%).
Time Frame: Pre-dose (within 60 minutes prior to dose), 0.5, 1, 2, 4, 6, anytime between 8 to 12 and 24 hours post-dose on Day 1
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percentage of drug concentration
Arm/Group | Talazoparib: Normal Hepatic Function | Talazoparib: Mild Hepatic Impairment | Talazoparib: Moderate Hepatic Impairment | Talazoparib: Severe Hepatic Impairment
Number analyzed (Participants) | 7 | 9 | 5 | 14
percentage of drug concentration | 28.76 (20) | 28.11 (14) | 27.47 (15) | 34.66 (17)

9. Secondary Outcome: Unbound Area Under the Free Plasma Concentration Time Curve From Zero to 24 Hours (AUC0-24u) of Talazoparib on Day 1
Description: AUC0-24u for unbound talazoparib was defined as the area under the free plasma concentration time curve from time 0 to 24 hours post-dose. AUC0-24u = fu*AUC0-24.
Time Frame: Pre-dose (within 60 minutes prior to dose), 0.5, 1, 2, 4, 6, anytime between 8 to 12 and 24 hours post-dose on Day 1
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter
Arm/Group | Talazoparib: Normal Hepatic Function | Talazoparib: Mild Hepatic Impairment | Talazoparib: Moderate Hepatic Impairment | Talazoparib: Severe Hepatic Impairment
Number analyzed (Participants) | 7 | 8 | 5 | 11
nanogram*hour per milliliter | 6.388 (42) | 7.569 (35) | 6.922 (14) | 7.528 (51)
Statistical Analysis 1: Comparison: Talazoparib: Normal Hepatic Function vs Talazoparib: Mild Hepatic Impairment; AUC0-24u was natural log-transformed and analyzed using ANOVA model with hepatic function group as a fixed effect; Test type: Other — Bioequivalence; Percent Ratio of Geometric Means = 118.47, 90% CI 2-sided [83.81 to 167.47]
Statistical Analysis 2: Comparison: Talazoparib: Normal Hepatic Function vs Talazoparib: Moderate Hepatic Impairment; AUC0-24u was natural log-transformed and analyzed using ANOVA model with hepatic function group as a fixed effect; Test type: Other — Bioequivalence; Percent Ratio of Geometric Means = 108.36, 90% CI 2-sided [73.25 to 160.30]
Statistical Analysis 3: Comparison: Talazoparib: Normal Hepatic Function vs Talazoparib: Severe Hepatic Impairment; AUC0-24u was natural log-transformed and analyzed using ANOVA model with hepatic function group as a fixed effect; Test type: Other — Bioequivalence; Percent Ratio of Geometric Means = 117.84, 90% CI 2-sided [85.29 to 162.83]

10. Secondary Outcome: Unbound Maximum Observed Plasma Concentration (Cmaxu) of Talazoparib on Day 1
Description: Cmaxu was defined as the maximum observed plasma concentration for unbound talazoparib. Cmaxu = fu*Cmax
Time Frame: Pre-dose (within 60 minutes prior to dose), 0.5, 1, 2, 4, 6, anytime between 8 to 12 and 24 hours post-dose on Day 1
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter
Arm/Group | Talazoparib: Normal Hepatic Function | Talazoparib: Mild Hepatic Impairment | Talazoparib: Moderate Hepatic Impairment | Talazoparib: Severe Hepatic Impairment
Number analyzed (Participants) | 7 | 8 | 5 | 13
nanogram per milliliter | 0.8823 (76) | 0.8345 (35) | 0.8131 (40) | 0.7448 (78)
Statistical Analysis 1: Comparison: Talazoparib: Normal Hepatic Function vs Talazoparib: Mild Hepatic Impairment; Cmaxu was natural log-transformed and analyzed using an ANOVA model with hepatic function group as a fixed effect; Test type: Other — Bioequivalence; Percent Ratio of Geometric Means = 94.58, 90% CI 2-sided [56.74 to 157.64]
Statistical Analysis 2: Comparison: Talazoparib: Normal Hepatic Function vs Talazoparib: Moderate Hepatic Impairment; Cmaxu was natural log-transformed and analyzed using an ANOVA model with hepatic function group as a fixed effect; Test type: Other — Bioequivalence; Percent Ratio of Geometric Means = 92.15, 90% CI 2-sided [51.69 to 164.26]
Statistical Analysis 3: Comparison: Talazoparib: Normal Hepatic Function vs Talazoparib: Severe Hepatic Impairment; Cmaxu was natural log-transformed and analyzed using an ANOVA model with hepatic function group as a fixed effect; Test type: Other — Bioequivalence; Percent Ratio of Geometric Means = 84.42, 90% CI 2-sided [53.14 to 134.10]

11. Secondary Outcome: Plasma Trough Concentration (Ctrough) of Talazoparib on Day 8, 15 and 22
Description: Ctrough was defined as plasma trough (pre-dose) concentration of talazoparib. Acceptance criteria for Ctrough on Day 15 and Day 22: received 10 consecutive days of dosing immediately before PK sampling day; Sample drawn within 24 +/-2 hours of the previous dose, and not more than +10 minute after the drug administration on the PK collection day. Ctrough on Day 8: received 7 consecutive days of dosing immediately before PK sampling day; sample drawn within 24 +/- 2 hours of the previous dose, and not more than +10 minute after the drug administration on the PK collection day.
Time Frame: Pre-dose on Day 8, 15 and 22
Population: Analysis population for this outcome measure included those participants who met acceptance criteria for Ctrough. Here 'number analyzed' signifies number of participants evaluable for each specified row.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter
Arm/Group | Talazoparib: Normal Hepatic Function | Talazoparib: Mild Hepatic Impairment | Talazoparib: Moderate Hepatic Impairment | Talazoparib: Severe Hepatic Impairment
Number analyzed (Participants) | 6 | 6 | 5 | 4
nanogram per milliliter
  Day 8: number analyzed (Participants) | 5 | 6 | 5 | 4
  Day 8 | 2.244 (22) | 4.807 (93) | 3.788 (80) | 3.329 (57)
  Day 15: number analyzed (Participants) | 6 | 2 | 3 | 4
  Day 15 | 2.857 (39) | NA (NA) — Data is not reported, as it was planned to report statistics when there were >=3 evaluable participants. | 2.909 (3) | 4.208 (86)
  Day 22: number analyzed (Participants) | 6 | 3 | 3 | 2
  Day 22 | 2.624 (28) | 3.699 (197) | 3.553 (8) | NA (NA) — Data is not reported, as it was planned to report statistics when there were >=3 evaluable participants.

12. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) of Talazoparib on Day 22
Description: Tmax was defined as the time to reach maximum observed plasma concentration of talazoparib.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Median (Full Range); unit: hour
Arm/Group | Talazoparib: Normal Hepatic Function | Talazoparib: Mild Hepatic Impairment | Talazoparib: Moderate Hepatic Impairment | Talazoparib: Severe Hepatic Impairment
Number analyzed (Participants) | 6 | 6 | 3 | 2
hour | 1.50 [0.50 to 2.13] | 2.13 [1.05 to 4.00] | 1.05 [1.00 to 2.75] | NA [NA to NA] — Data is not reported, as it was planned to report statistics when there were >=3 evaluable participants.

13. Secondary Outcome: Fraction of Unbound (fu) Plasma Talazoparib on Day 22
Description: as for outcome 8
Time Frame: as for outcome 1
Population: Analysis population included participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percentage of drug concentration
Arm/Group | Talazoparib: Normal Hepatic Function | Talazoparib: Mild Hepatic Impairment | Talazoparib: Moderate Hepatic Impairment | Talazoparib: Severe Hepatic Impairment
Number analyzed (Participants) | 6 | 8 | 3 | 5
percentage of drug concentration | 26.98 (23) | 27.71 (18) | 27.10 (9) | 33.92 (25)

14. Secondary Outcome: Accumulation Ratio (Rac) of Plasma Talazoparib
Description: Accumulation ratio for AUC0-24 was calculated as area under the curve from time zero to 24 hours on Day 22 divided by area under the curve from time zero to 24 hours on Day 1.
Time Frame: Pre-dose (within 60 minutes prior to dose) on Day 1, pre-dose(24 hours +/- 60 minutes from the previous dose on Day 21 but within 60 minutes prior to next dose) on Day 22 and 0.5, 1, 2, 4, 6, anytime between 8 to 12 and 24 hours post-dose on Days 1 and 22
Population: PK evaluable analysis population was analyzed. Here, "Overall Number of Participants Analyzed" =participants evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Talazoparib: Normal Hepatic Function | Talazoparib: Mild Hepatic Impairment | Talazoparib: Moderate Hepatic Impairment | Talazoparib: Severe Hepatic Impairment
Number analyzed (Participants) | 6 | 5 | 3 | 1
ratio | 5.070 (24) | 5.134 (68) | 4.771 (31) | NA (NA) — Data is not reported, as it was planned to report statistics when there were >=3 evaluable participants.

15. Secondary Outcome: Apparent Clearance (CL/F) of Plasma Talazoparib on Day 22
Description: Talazoparib clearance is a measure of the rate at which talazoparib is metabolized or eliminated by normal biological processes.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter per hour
Arm/Group | Talazoparib: Normal Hepatic Function | Talazoparib: Mild Hepatic Impairment | Talazoparib: Moderate Hepatic Impairment | Talazoparib: Severe Hepatic Impairment
Number analyzed (Participants) | 6 | 6 | 3 | 2
liter per hour | 5.070 (24) | 5.134 (68) | 4.771 (31) | NA (NA) — Data is not reported, as it was planned to report statistics when there were >=3 evaluable participants.

16. Secondary Outcome: Unbound Apparent Clearance (CLu/F) of PlasmaTalazoparib on Day 22
Description: Clearance of unbound talazoparib is a measure of the rate at which unbound talazoparib is metabolized or eliminated by normal biological processes.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter per hour
Arm/Group | Talazoparib: Normal Hepatic Function | Talazoparib: Mild Hepatic Impairment | Talazoparib: Moderate Hepatic Impairment | Talazoparib: Severe Hepatic Impairment
Number analyzed (Participants) | 6 | 6 | 3 | 2
liter per hour | 16.57 (11) | 11.09 (84) | 14.92 (35) | NA (NA) — Data is not reported, as it was planned to report statistics when there were >=3 evaluable participants.

17. Secondary Outcome: Amount of Talazoparib Excreted Unchanged in Urine From Time Zero to 24 Hours (Ae 0-24) on Day 1
Description: Ae 0-24 is the amount of talazoparib excreted unchanged in urine from time 0 to 24 hours post dose.
Time Frame: A single void at pre-dose, post-dose at any time between 0 to 12 and any time between 12 to 24 hours on Day 1
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milligram
Arm/Group | Talazoparib: Normal Hepatic Function | Talazoparib: Mild Hepatic Impairment | Talazoparib: Moderate Hepatic Impairment | Talazoparib: Severe Hepatic Impairment
Number analyzed (Participants) | 7 | 8 | 4 | 8
milligram | 0.03816 (79) | 0.03534 (71) | 0.04292 (85) | 0.02319 (107)

18. Secondary Outcome: Percentage of Talazoparib Excreted in Urine From Time Zero to 24 Hours (Ae 0-24%) on Day 1
Description: Ae0-24% was defined as the amount of talazoparib excreted in urine from time 0 to 24 hours expressed as percentage of administered dose.
Time Frame: A single void at pre-dose, post-dose at any time between 0 to 12 and any time between 12 to 24 hours on Day 1
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percentage of dose
Arm/Group | Talazoparib: Normal Hepatic Function | Talazoparib: Mild Hepatic Impairment | Talazoparib: Moderate Hepatic Impairment | Talazoparib: Severe Hepatic Impairment
Number analyzed (Participants) | 7 | 8 | 4 | 8
percentage of dose | 7.638 (79) | 7.070 (71) | 8.582 (85) | 4.641 (107)

19. Secondary Outcome: Amount of Talazoparib Excreted Unchanged in Urine From Time Zero to 24 Hours (Ae 0-24) on Day 22
Description: Ae 0-24 is the amount of talazoparib excreted unchanged in urine from time 0 to 24 hours post dose.
Time Frame: Urine voided post-dose at any time between 0 to 12 and any time between 12 to 24 hours on Day 22
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milligram
Arm/Group | Talazoparib: Normal Hepatic Function | Talazoparib: Mild Hepatic Impairment | Talazoparib: Moderate Hepatic Impairment | Talazoparib: Severe Hepatic Impairment
Number analyzed (Participants) | 6 | 5 | 3 | 2
milligram | 0.2229 (30) | 0.1819 (34) | 0.1867 (32) | NA (NA) — Data is not reported, as it was planned to report statistics when there were >=3 evaluable participants.

20. Secondary Outcome: Percentage of Talazoparib Excreted in Urine From Time 0 to 24 Hours (Ae 0-24%) on Day 22
Description: Ae 0-24% was defined as the amount of talazoparib excreted in urine from time 0 to 24 hours expressed as percentage of administered dose.
Time Frame: Urine voided post-dose at any time between 0 to 12 and any time between 12 to 24 hours (hrs) on Day 22
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percentage of dose
Arm/Group | Talazoparib: Normal Hepatic Function | Talazoparib: Mild Hepatic Impairment | Talazoparib: Moderate Hepatic Impairment | Talazoparib: Severe Hepatic Impairment
Number analyzed (Participants) | 6 | 5 | 3 | 2
percentage of dose | 44.58 (30) | 36.36 (34) | 37.40 (31) | NA (NA) — Data is not reported, as it was planned to report statistics when there were >=3 evaluable participants.

21. Secondary Outcome: Renal Clearance (CLr) of Talazoparib on Day 22
Description: Renal clearance was calculated as cumulative amount of drug excreted in urine during the 24 hours dosing interval (Ae) divided by area under the plasma concentration time-curve from time zero to 24 hours post dose (AUC0-24).
Time Frame: Ae: Post-dose at any time between 0 to 12, 12 to 24 hrs on Day 22; AUC0-24: Pre-dose (24 hrs +/- 60 minutes from previous dose on Day 21 but within 60 minutes prior to next dose), 0.5, 1, 2, 4, 6, any time between 8 to12, 24 hrs post-dose on Day 22
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters per hour
Arm/Group | Talazoparib: Normal Hepatic Function | Talazoparib: Mild Hepatic Impairment | Talazoparib: Moderate Hepatic Impairment | Talazoparib: Severe Hepatic Impairment
Number analyzed (Participants) | 6 | 5 | 3 | 2
liters per hour | 1.993 (57) | 1.449 (92) | 1.510 (39) | NA (NA) — Data is not reported, as it was planned to report statistics when there were >=3 evaluable participants.

22. Other Pre Specified Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received investigational product without regard to possibility of causal relationship. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly; medically important events. TEAEs were events between first dose of Talazoparib and up to 30 days after the last dose of Talazoparib (up to 52 days) that were absent before treatment or that worsened relative to pretreatment state. AEs included both SAEs and all non-SAEs.
Time Frame: Baseline up to 30 days after last dose of study drug (up to 52 days)
Population: Safety analysis set included all participants who received any amount of talazoparib.
Measure: Count of Participants; unit: Participants
Arm/Group | Talazoparib: Normal Hepatic Function | Talazoparib: Mild Hepatic Impairment | Talazoparib: Moderate Hepatic Impairment | Talazoparib: Severe Hepatic Impairment
Number analyzed (Participants) | 7 | 10 | 5 | 16
Participants
  TEAEs | 6 | 8 | 3 | 14
  SAEs | 1 | 3 | 2 | 13

23. Other Pre Specified Outcome: Number of Participants With TEAEs Leading to Study Drug Discontinuation
Description: An AE was any untoward medical occurrence in a participant who received investigational product without regard to possibility of causal relationship. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly; medically important events. Treatment-emergent were events between first dose of Talazoparib and up to 30 days after the last dose of Talazoparib (up to 52 days) that were absent before treatment or that worsened relative to pretreatment state. AEs included both SAEs and non-SAEs. Number of participants with TEAEs leading to study drug discontinuation are reported.
Time Frame: Baseline up to 30 days after last dose of study drug (up to 52 days)
Population: Safety analysis set included all participants who received any amount of talazoparib.
Measure: Count of Participants; unit: Participants
Arm/Group | Talazoparib: Normal Hepatic Function | Talazoparib: Mild Hepatic Impairment | Talazoparib: Moderate Hepatic Impairment | Talazoparib: Severe Hepatic Impairment
Number analyzed (Participants) | 7 | 10 | 5 | 16
Participants | 0 | 2 | 2 | 12

24. Other Pre Specified Outcome: Number of Participants With TEAEs Resulting in Death
Description: An AE was any untoward medical occurrence in a participant who received investigational product without regard to possibility of causal relationship. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly; medically important events. Treatment-emergent were events between first dose of Talazoparib and up to 30 days after the last dose of Talazoparib (up to 52 days) that were absent before treatment or that worsened relative to pretreatment state. AEs included both SAEs and non-SAEs. Number of participants with TEAEs resulting in death are reported.
Time Frame: Baseline up to 30 days after last dose of study drug (up to 52 days)
Population: Safety analysis set included all participants who received any amount of talazoparib.
Measure: Count of Participants; unit: Participants
Arm/Group | Talazoparib: Normal Hepatic Function | Talazoparib: Mild Hepatic Impairment | Talazoparib: Moderate Hepatic Impairment | Talazoparib: Severe Hepatic Impairment
Number analyzed (Participants) | 7 | 10 | 5 | 16
Participants | 0 | 0 | 1 | 7

25. Other Pre Specified Outcome: Number of Participants With Treatment Emergent Treatment Related Adverse Events and SAEs
Description: A treatment-related adverse event was any untoward medical occurrence attributed to talazoparib in a participant who received talazoparib. A treatment-related serious adverse event was a treatment-related adverse event resulting in any of the following outcomes or deemed significant for any other reason: death; life-threatening experience (immediate risk of dying); initial or prolonged inpatient hospitalization; persistent or significant disability/incapacity; Congenital anomaly. Relatedness to talazoparib was assessed by the investigator.
Time Frame: Baseline up to 30 days after last dose of study drug (up to 52 days)
Population: Safety analysis set included all participants who received any amount of talazoparib.
Measure: Count of Participants; unit: Participants
Arm/Group | Talazoparib: Normal Hepatic Function | Talazoparib: Mild Hepatic Impairment | Talazoparib: Moderate Hepatic Impairment | Talazoparib: Severe Hepatic Impairment
Number analyzed (Participants) | 7 | 10 | 5 | 16
Participants
  AEs | 4 | 3 | 0 | 2
  SAEs | 0 | 0 | 0 | 0

26. Secondary Outcome: Number of Participants With Clinically Significant Laboratory Abnormalities
Description: Clinically significant laboratory abnormalities included aspartate transaminase (AST) or alanine aminotransferase (ALT) >=3 times ULN (>5 *ULN if baseline ALT/AST is >3 *ULN) and total bilirubin (TBL) >2 times ULN or INR >1.5, AST or ALT >=3 times ULN with signs and symptoms consistent with hepatitis and/or eosinophilia (>=500 eosinophils/microliter).
Time Frame: Baseline up to 30 days after last dose of study drug (up to 52 days)
Population: Safety analysis set included all participants who received any amount of talazoparib.
Measure: Count of Participants; unit: Participants
Arm/Group | Talazoparib: Normal Hepatic Function | Talazoparib: Mild Hepatic Impairment | Talazoparib: Moderate Hepatic Impairment | Talazoparib: Severe Hepatic Impairment
Number analyzed (Participants) | 7 | 10 | 5 | 16
Participants | 0 | 0 | 0 | 3

27. Secondary Outcome: Change From Baseline in Vital Sign -Blood Pressure at Day 2, 8, 15, 22 and End of Study
Description: Systolic blood pressure and diastolic blood pressure were evaluated for examination of vital signs.
Time Frame: Baseline, Day 2, 8, 15, 22 and End of Study (Day 52)
Population: Safety analysis set included all participants who received any amount of talazoparib. Here, 'number analyzed' signifies participants evaluable for each specified row.
Measure: Mean (Standard Deviation); unit: millimeter of mercury (mmHg)
Arm/Group | Talazoparib: Normal Hepatic Function | Talazoparib: Mild Hepatic Impairment | Talazoparib: Moderate Hepatic Impairment | Talazoparib: Severe Hepatic Impairment
Number analyzed (Participants) | 7 | 10 | 5 | 16
millimeter of mercury (mmHg)
  Systolic Blood Pressure: Baseline | 128.1 (19.22) | 110.3 (11.84) | 121.8 (23.15) | 115.8 (13.57)
  Systolic Blood Pressure: Change at Day 2: number analyzed (Participants) | 7 | 7 | 4 | 13
  Systolic Blood Pressure: Change at Day 2 | -12.3 (17.72) | -1.1 (12.86) | -12.5 (14.48) | 2.2 (10.43)
  Systolic Blood Pressure: Change at Day 8: number analyzed (Participants) | 7 | 8 | 5 | 12
  Systolic Blood Pressure: Change at Day 8 | -2.0 (20.22) | -2.8 (9.85) | -5.6 (11.97) | -5.3 (10.80)
  Systolic Blood Pressure: Change at Day 15: number analyzed (Participants) | 7 | 8 | 4 | 8
  Systolic Blood Pressure: Change at Day 15 | -8.4 (8.64) | 0.3 (12.08) | -6.0 (23.47) | -2.3 (13.91)
  Systolic Blood Pressure: Change at Day 22: number analyzed (Participants) | 6 | 8 | 3 | 9
  Systolic Blood Pressure: Change at Day 22 | -7.5 (15.10) | -4.3 (14.30) | -10.7 (32.56) | -7.8 (17.20)
  Systolic Blood Pressure: Change at end of study (Day 52): number analyzed (Participants) | 4 | 7 | 0 | 1
  Systolic Blood Pressure: Change at end of study (Day 52) | -0.8 (18.36) | 0.7 (14.22) |  | -26.0
  Diastolic Blood Pressure: Baseline | 75.9 (12.52) | 65.9 (10.77) | 68.4 (5.59) | 73.9 (10.60)
  Diastolic Blood Pressure: Change at Day 2: number analyzed (Participants) | 7 | 7 | 4 | 13
  Diastolic Blood Pressure: Change at Day 2 | -5.0 (6.76) | 4.1 (7.69) | -4.5 (6.19) | -0.8 (7.03)
  Diastolic Blood Pressure: Change at Day 8: number analyzed (Participants) | 7 | 8 | 5 | 12
  Diastolic Blood Pressure: Change at Day 8 | -1.0 (12.04) | 4.1 (6.66) | -0.8 (9.12) | -4.1 (9.91)
  Diastolic Blood Pressure: Change at Day 15: number analyzed (Participants) | 7 | 8 | 4 | 8
  Diastolic Blood Pressure: Change at Day 15 | -1.4 (6.92) | 0.9 (9.00) | 0.8 (10.84) | -2.1 (4.97)
  Diastolic Blood Pressure: Change at Day 22: number analyzed (Participants) | 6 | 8 | 3 | 9
  Diastolic Blood Pressure: Change at Day 22 | -3.5 (9.14) | -3.0 (7.82) | -3.3 (15.53) | -6.0 (11.17)
  Diastolic Blood Pressure: Change at end of study (Day 52): number analyzed (Participants) | 4 | 7 | 0 | 1
  Diastolic Blood Pressure: Change at end of study (Day 52) | -0.3 (8.26) | 1.9 (7.52) |  | -17.0

28. Secondary Outcome: Change From Baseline in Vital Sign- Heart Rate at Day 2, 8, 15, 22 and End of Study
Description: Heart rate was measured in beats per minute.
Time Frame: Baseline, Day 2, 8, 15, 22 and End of Study (Day 52)
Population: as for outcome 27
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Talazoparib: Normal Hepatic Function | Talazoparib: Mild Hepatic Impairment | Talazoparib: Moderate Hepatic Impairment | Talazoparib: Severe Hepatic Impairment
Number analyzed (Participants) | 7 | 10 | 5 | 16
beats per minute
  Baseline | 75.9 (7.67) | 89.2 (19.34) | 87.4 (22.13) | 92.3 (16.76)
  Change at Day 2: number analyzed (Participants) | 7 | 7 | 4 | 13
  Change at Day 2 | 3.0 (7.64) | 4.7 (10.01) | 1.0 (6.16) | 1.4 (11.01)
  Change at Day 8: number analyzed (Participants) | 7 | 8 | 5 | 12
  Change at Day 8 | 1.7 (7.78) | 3.5 (16.10) | 1.6 (4.67) | -2.7 (8.79)
  Change at Day 15: number analyzed (Participants) | 7 | 8 | 4 | 8
  Change at Day 15 | 5.1 (9.82) | -6.0 (12.76) | 2.5 (7.05) | 3.8 (15.52)
  Change at Day 22: number analyzed (Participants) | 6 | 8 | 3 | 9
  Change at Day 22 | 2.2 (9.81) | -9.9 (20.38) | -2.0 (1.00) | 2.3 (19.16)
  Change at end of study (Day 52): number analyzed (Participants) | 4 | 7 | 0 | 1
  Change at end of study (Day 52) | 8.5 (11.90) | 3.1 (15.56) |  | 23.0

29. Secondary Outcome: Change From Baseline in Vital Sign- Respiratory Rate at Day 8, 15, 22 and End of Study
Description: Respiratory rate was measured in terms of breaths per minute.
Time Frame: Baseline, Day 8, 15, 22 and End of Study (Day 52)
Population: as for outcome 27
Measure: Mean (Standard Deviation); unit: breaths per minute
Arm/Group | Talazoparib: Normal Hepatic Function | Talazoparib: Mild Hepatic Impairment | Talazoparib: Moderate Hepatic Impairment | Talazoparib: Severe Hepatic Impairment
Number analyzed (Participants) | 7 | 10 | 5 | 16
breaths per minute
  Baseline | 18.3 (2.63) | 17.1 (1.20) | 16.8 (0.84) | 17.4 (1.63)
  Change at Day 8: number analyzed (Participants) | 7 | 8 | 5 | 12
  Change at Day 8 | -0.3 (2.06) | 0.6 (1.77) | 1.2 (2.39) | -0.1 (2.19)
  Change at Day 15: number analyzed (Participants) | 7 | 8 | 3 | 8
  Change at Day 15 | -1.6 (3.15) | -0.4 (1.51) | 0.3 (1.53) | 0.4 (1.51)
  Change at Day 22: number analyzed (Participants) | 6 | 8 | 3 | 9
  Change at Day 22 | -0.2 (0.98) | -0.6 (1.41) | 1.3 (0.58) | 1.1 (1.17)
  Change at end of study (Day 52): number analyzed (Participants) | 4 | 7 | 0 | 1
  Change at end of study (Day 52) | -0.5 (1.00) | 0.1 (1.46) |  | 2.0

30. Secondary Outcome: Change From Baseline in Vital Sign- Weight at Day 8, 15, 22 and End of Study
Time Frame: Baseline, Day 8, 15, 22 and End of Study (Day 52)
Population: as for outcome 27
Measure: Mean (Standard Deviation); unit: kilogram
Arm/Group | Talazoparib: Normal Hepatic Function | Talazoparib: Mild Hepatic Impairment | Talazoparib: Moderate Hepatic Impairment | Talazoparib: Severe Hepatic Impairment
Number analyzed (Participants) | 7 | 10 | 5 | 16
kilogram
  Baseline | 82.01 (15.749) | 63.07 (11.493) | 77.78 (17.070) | 66.98 (12.979)
  Change at Day 8: number analyzed (Participants) | 7 | 8 | 5 | 12
  Change at Day 8 | -0.04 (0.943) | -0.10 (1.865) | -2.02 (1.656) | -1.50 (3.728)
  Change at Day 15: number analyzed (Participants) | 7 | 8 | 4 | 8
  Change at Day 15 | -0.36 (0.621) | -0.09 (2.119) | -1.78 (0.900) | -1.29 (5.025)
  Change at Day 22: number analyzed (Participants) | 6 | 8 | 3 | 9
  Change at Day 22 | -0.78 (0.546) | 0.28 (1.647) | -1.57 (0.462) | -2.06 (5.416)
  Change at end of study (Day 52): number analyzed (Participants) | 4 | 7 | 0 | 1
  Change at end of study (Day 52) | 0.48 (1.839) | 1.81 (1.577) |  | 0.90

31. Secondary Outcome: Number of Participants Who Met the Pre-specified 12-Lead Electrocardiogram (ECG) Criteria
Description: Pre-specified 12-Lead electrocardiogram (ECG) Criteria: QTCF (Fridericia's correction formula) : >=450 to <480 milliseconds, >=480 to <500 milliseconds, >=500 milliseconds, increase from baseline >=30 - <60, increase from baseline >=60, PR interval: >=300 milliseconds, increase from baseline >=25%; QRS duration: >=140 milliseconds, increase from baseline >=50%; QT interval: >=500 milliseconds; QT Interval: >= 500 milliseconds.
Time Frame: Baseline up to 30 days after last dose of study drug (up to 52 days)
Population: Safety analysis set included all participants who received any amount of talazoparib.
Measure: Count of Participants; unit: Participants
Arm/Group | Talazoparib: Normal Hepatic Function | Talazoparib: Mild Hepatic Impairment | Talazoparib: Moderate Hepatic Impairment | Talazoparib: Severe Hepatic Impairment
Number analyzed (Participants) | 7 | 10 | 5 | 16
Participants
  QTCF: >=450 - <480 milliseconds | 2 | 2 | 1 | 4
  QTCF: >=480 - <500 milliseconds | 0 | 0 | 0 | 1
  QTCF: >=500 milliseconds | 0 | 0 | 0 | 1
  QTCF: Increase from baseline >=30 - <60 milliseconds | 2 | 0 | 0 | 3
  QTCF: Increase from baseline >=60 milliseconds | 0 | 1 | 0 | 1
  PR Interval: >=300 milliseconds | 1 | 0 | 0 | 0
  PR Interval: Increase from baseline >=25% | 1 | 0 | 0 | 2
  QRS Duration: >=140 milliseconds | 0 | 0 | 0 | 1
  QRS Duration: Increase from baseline >=50% | 0 | 0 | 0 | 0
  QT Interval: >=500 milliseconds | 0 | 0 | 1 | 0

32. Secondary Outcome: Number of Participants With Eastern Cooperative Oncology Group (ECOG) Performance Status
Description: As per ECOG, participant's performance status was measured as: 0=fully active/able to carry on all pre-disease activities without restriction; 1= restricted in physically strenuous activity but ambulatory and able to carry out work of a light and sedentary nature, e.g., light housework, office work; 2= ambulatory and capable of all self-care, but unable to carry out any work activities, up and about more than 50% of waking hours; 3=capable of only limited self-care, confined to bed/chair >50% of waking hours; 4=completely disabled, cannot carry on any self-care, totally confined to bed/chair.
Time Frame: Screening (2 to 28 days prior to Day 1), Day -1 (1 day prior to Day 1), safety follow up (Visit up to Day 52)
Population: as for outcome 27
Measure: Count of Participants; unit: Participants
Arm/Group | Talazoparib: Normal Hepatic Function | Talazoparib: Mild Hepatic Impairment | Talazoparib: Moderate Hepatic Impairment | Talazoparib: Severe Hepatic Impairment
Number analyzed (Participants) | 7 | 10 | 5 | 16
Participants
  Screening: ECOG Performance Status: 0 | 3 | 1 | 1 | 0
  Screening: ECOG Performance Status: 1 | 4 | 8 | 2 | 12
  Screening: ECOG Performance Status: 2 | 0 | 1 | 2 | 4
  Screening: ECOG Performance Status: 3 | 0 | 0 | 0 | 0
  Screening: ECOG Performance Status: 4 | 0 | 0 | 0 | 0
  Day -1: number analyzed (Participants) | 7 | 10 | 4 | 15
  Day -1: ECOG Performance Status: 0 | 2 | 0 | 0 | 0
  Day -1: ECOG Performance Status: 1 | 5 | 9 | 2 | 11
  Day -1: ECOG Performance Status: 2 | 0 | 1 | 2 | 4
  Day -1: ECOG Performance Status: 3 | 0 | 0 | 0 | 0
  Day -1: ECOG Performance Status: 4 | 0 | 0 | 0 | 0
  Safety follow up: number analyzed (Participants) | 4 | 6 | 0 | 1
  Safety follow up: ECOG Performance Status: 0 | 2 | 1 | 0 | 0
  Safety follow up: ECOG Performance Status: 1 | 2 | 4 | 0 | 1
  Safety follow up: ECOG Performance Status: 2 | 0 | 1 | 0 | 0
  Safety follow up: ECOG Performance Status: 3 | 0 | 0 | 0 | 0
  Safety follow up: ECOG Performance Status: 4 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline up to 30 days after last dose of study drug (up to 52 days)
Description: Same event may appear as AE and SAE, what is presented are distinct events. Event may be categorized as serious in 1 participant and as non-serious in another participant or 1 participant may have experienced both serious and non-serious event during study.
Arm/Group | Talazoparib: Normal Hepatic Function | Talazoparib: Mild Hepatic Impairment | Talazoparib: Moderate Hepatic Impairment | Talazoparib: Severe Hepatic Impairment
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/10 | 1/5 | 7/16
Serious Adverse Events (participants affected / at risk) | 1/7 | 3/10 | 2/5 | 13/16
Other Adverse Events (participants affected / at risk) | 6/7 | 7/10 | 3/5 | 10/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Talazoparib: Normal Hepatic Function (N=7) | Talazoparib: Mild Hepatic Impairment (N=10) | Talazoparib: Moderate Hepatic Impairment (N=5) | Talazoparib: Severe Hepatic Impairment (N=16)
Disease progression (General disorders) | 0 | 0 | 0 | 4
Pyrexia (General disorders) | 0 | 1 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 1 | 2
Cholangitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 3
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 2
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 2
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Hepatic encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 2
Facial paralysis (Nervous system disorders) | 0 | 1 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 0 | 0 | 0 | 1
Coronary artery occlusion (Cardiac disorders) | 0 | 1 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Talazoparib: Normal Hepatic Function (N=7) | Talazoparib: Mild Hepatic Impairment (N=10) | Talazoparib: Moderate Hepatic Impairment (N=5) | Talazoparib: Severe Hepatic Impairment (N=16)
Fatigue (General disorders) | 4 | 1 | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 2 | 1 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 2 | 0 | 3
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 2 | 1 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 2
Hepatic encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 2
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Coagulopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2
Constipation (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 2
Oedema peripheral (General disorders) | 0 | 0 | 0 | 2
Sepsis (Infections and infestations) | 0 | 0 | 0 | 2
Breast pain (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Chills (General disorders) | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Device related infection (Infections and infestations) | 0 | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Ammonia increased (Investigations) | 0 | 0 | 0 | 1
Cholangitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Device occlusion (Product Issues) | 0 | 0 | 0 | 1
Generalised oedema (General disorders) | 0 | 0 | 0 | 1
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Haematoma (Vascular disorders) | 0 | 0 | 0 | 1
Hepatosplenomegaly (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2018-09-14): https://cdn.clinicaltrials.gov/large-docs/76/NCT02997176/Prot_000.pdf
  • Statistical Analysis Plan (2019-12-09): https://cdn.clinicaltrials.gov/large-docs/76/NCT02997176/SAP_001.pdf